CLINICAL TRIAL: NCT04744025
Title: A Double-blind Prospective Randomized Clinical Trial Comparing Euploidy Rates Among Embryos Created From Sibling Oocytes Injected With Sperm Processed by Microfluidics or by Density Gradient Centrifugation
Brief Title: Microfluidics Versus Gradient Centrifugation Effect on Euploidy Rates
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lawrence Engmann (Other)
Collaborators: The Center for Advanced Reproductive Services, P.C. (Other); ZyMot Fertility (Unknown)
Responsible Party: Sponsor-Investigator, Lawrence Engmann, Principal Investigator, The Center for Advanced Reproductive Services, P.C.
Organization: UConn Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-106R-1
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Infertility; Recurrent Pregnancy Loss
Keywords: Microfluidics; Density gradient centrifugation; In vitro fertilization; Preimplantation genetic testing; Euploidy; Sperm processing
MeSH Terms: conditions — Infertility | interventions — Centrifugation, Density Gradient

STUDY DESIGN:
Intervention Model Description: Sibling oocyte study: Participants will have their oocytes (eggs) divided into two groups. Half of the eggs will be injected with sperm processed in the normal way, and half will be injected with sperm processed via a microfluidics chamber.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, clinical providers, investigators and Outcome assessors will be blinded to outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Microfluidics (Experimental): Half of participants eggs will be injected with sperm processed using a microfluidics chamber.
  Interventions: Device: Microfluidics chamber
- Density gradient centrifugation (Active Comparator): Half of participants eggs will be injected with sperm processed using a density gradient centrifugation (the standard method).
  Interventions: Other: Density Gradient Centrifugation

INTERVENTIONS:
Device: Microfluidics chamber — Unwashed sperm will be placed into the inlet chamber of the microfluidics device. The most motile sperm will swim to the outlet chamber, and these sperms will be used for intracytoplasmic sperm injection (ICSI) into the eggs.
  Other Names: ZyMot Fertility (device brand name)
  Arms: Microfluidics
Other: Density Gradient Centrifugation — Sperm will be washed and centrifuged according to standard protocol, and these washed sperm will be used for ICSI.
  Arms: Density gradient centrifugation

SUMMARY:
This research is being done to determine if using a microfluidics chamber, a device used to process sperm, will be effective in improving the rates of embryos with normal chromosomes (structures that carry genetic information) during in vitro fertilization (IVF) treatment. The investigators hypothesize that this device is effective at improving rates of normal chromosomes among embryos.

DETAILED DESCRIPTION:
As part of the in vitro fertilization (IVF) process, eggs are removed from the ovaries and are inseminated (mixed) or injected with sperm. In order for fertilization to occur, the sperm cells must be separated from the semen before introducing them to the eggs. Currently, sperm are isolated from the semen using a series of wash steps in a centrifuge (device to spin and concentrate the sperm). This requires processing at high speeds in order to separate motile sperm from the other parts of the semen. Although it is common practice, it is possible that this method of processing the semen may cause damage to the sperm cells.

Alternatively, a microfluidics chamber can be used to choose the best sperm. A microfluidics chamber is a small device in which the unwashed sperm can be placed at one end. Sperm that are moving forward will swim through the chamber and come out the other end. Dead sperm are left behind and the sperm with the best motility (how normally they move forward) and normal morphology (how the sperm looks) will make it to the other end of the chamber. These sperm can then be chosen for injection into the egg. This device is FDA-approved for this purpose and is commercially available and is currently routinely used in the IVF lab utilized by the investigators as well as most labs in the country.

Some small initial studies showed that a higher number of embryos with higher quality were made with sperm selected from a microfluidics chamber. In another recent study, the chances of creating an embryo with a normal number of chromosomes (structures that carry genetic information) was also slightly higher if a microfluidics chamber was used to process the sperm. This might be because sperm that have the highest motility and normal morphology may also be more likely to be genetically normal. However, there are no good-quality studies looking at the rates of embryos with normal chromosomes created from using a microfluidics chamber to process sperm.

The purpose of this research study is to determine whether using a microfluidics chamber to process sperm for injection into eggs increases the rates of embryos with normal chromosomes. At the time of egg retrieval, participants will have their eggs randomized (like the flip of a coin) into two groups. Half of the eggs will be injected with sperm processed using gradient centrifugation, the standard method. The other half of the eggs will be injected with sperm processed using a microfluidics chamber. The goal is to determine the rate of embryos with normal chromosomes in each group. Other goals include looking at how many embryos develop to good quality blastocysts and are biopsied and how many patients get pregnant after embryo transfer.

ELIGIBILITY:
Inclusion criteria:

* Subjects are nonpregnant females ≥ 18 years and ≤ 42 years of age.
* Subjects obtain ≥ 6 mature oocytes at the time of oocyte retrieval or at the time of ICSI.
* Subjects are utilizing ICSI for fertilization.
* Subjects are utilizing PGT-A (PGT for aneuploidy).
* Subjects are able to understand, read, and write in English at a fifth-grade level.
* Subjects are willing to comply with study protocol and procedures and provide written informed consent.

Exclusion criteria:

* Subjects are utilizing donor oocytes, donor sperm, or gestational carrier.
* Subjects have a diagnosis of severe male factor infertility (sperm concentration < 5 mil/mL at semen analysis).
* Subjects are utilizing surgically removed sperm (e.g. via testicular sperm aspiration [TESA] or microsurgical epididymal sperm aspiration [MESA]).
* Subjects are utilizing frozen/thawed sperm.
* Subjects are utilizing frozen/thawed oocytes.
* Subjects are undergoing a day 3 (cleavage stage) embryo transfer.
* Subjects obtain < 6 mature oocytes at the time of oocyte retrieval or at the time of ICSI.
* Subjects obtain ≥ 6 mature oocytes but choose to fertilize fewer than 6 of them.
* Sperm sample parameters are low on the day of oocyte retrieval (semen volume < 1.0 mL or concentration < 1 million motile/mL).
* Male partner has an infectious disease.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Nonpregnant females underoing in vitro fertilization (IVF) with intracytoplasmic sperm injection (ICSI) and preimplantation genetic testing (PGT)
Enrollment: 150 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Euploidy rate of resulting embryos | Within 2-4 weeks of IVF cycle
  Rate of embryos with normal chromosomes in both groups

SECONDARY OUTCOMES:
Pregnancy rates after transfer of euploid embryos | Within 1-2 cycles of fresh IVF cycle
  Pregnancy rate after one euploid embryo (from either experimental or control group) is transferred back into the participant in a subsequent cycle

OTHER OUTCOMES:
DNA fragmentation results | 1-2 years after initial study completed
  Compare DNA fragmentation results between groups

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Engmann, MD, Principal Investigator — UConn Health; Alison Bartolucci, PhD, Principal Investigator — The Center for Advanced Reproductive Services, P.C.
Locations (1):
- The Center for Advanced Reproductive Services, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at this time, may be available upon request in the future

REFERENCES:
- [Derived] Godiwala P, Kwieraga J, Almanza E, Neuber E, Grow D, Benadiva C, Makhijani R, DiLuigi A, Schmidt D, Bartolucci A, Engmann L. The impact of microfluidics sperm processing on blastocyst euploidy rates compared with density gradient centrifugation: a sibling oocyte double-blinded prospective randomized clinical trial. Fertil Steril. 2024 Jul;122(1):85-94. doi: 10.1016/j.fertnstert.2024.02.021. Epub 2024 Feb 15. PMID 38367686
- See also: The Center for Advanced Reproductive Services Website — https://www.uconnfertility.com/